#### **Research Information Sheet**

Title of Study: Testing a Novel Instagram Intervention for Alcohol Use – Main Study

Principal Investigator (PI): Halle Thomas

Department of Psychology halle.a.thomas@wayne.edu

#### Introduction:

You are being asked to participate in a research study. The purpose of this form is to provide you information that may affect your decision as to whether or not to participate. Your participation is <u>entirely voluntary</u>, and you can refuse to participate at any time without penalty.

## What is this study about & why is it being done?

You are being asked to participate in a research study about social media and alcohol use because you are a Prolific user who has completed our screening survey and has indicated that you have used alcohol recently and regularly use Instagram. This study is being conducted at Wayne State University. The purpose of this form is to provide you information to decide whether or not to you want to participate in this research study. Your participation is <u>entirely voluntary</u>, and you can refuse to participate or withdraw at any time without penalty.

A description of this clinical trial will be available on http://ClinicalTrials.gov as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## What Will I Do and How Long Will It Take?

If you take part in the study, you will be asked to complete a 20-minute baseline survey, which will ask about demographic information, your alcohol use, and mood.

If randomly assigned to take part in the novel intervention, you will be given the study username and URL and will be asked to request to follow the page as soon as possible. You will also be asked to provide your own Instagram URL/username. Once the page begins posting content, you will be expected to 'like' posts as they appear on your newsfeed and to interact with the content as much as feels comfortable.

All participants, including those not assigned to take part in the intervention, will gain access to a follow-up survey ten weeks after the start of the intervention. This survey will require another 20-30 minutes to complete. You have the option of skipping any questions that you do not want to answer. Your name will not be attached to any of your answers, and your data will be kept confidential. The entire study will be completed in three months following the start of the intervention.

## What are the Possible Benefits of participating in this study?

This study is not designed with a direct benefit to participants; however, information from this study may benefit other people now or in the future.

#### What are the risks and discomforts of participating in this study?

The risks to participating in this study are similar to risks encountered in everyday life. These risks include:

02/13/2024 - 02/12/2027 APPROVAL PERIOD

WAYNE STATE UNIVERSITY
INSTITUTIONAL REVIEW BOARD

IRB-23-11-6344

Form Date: 12/2023

- Some questions may be personal or upsetting. You do not need to answer any questions that do not want to answer.
- Possible loss of confidentiality: there is a chance your data could be seen by someone who shouldn't have access to it. We're minimizing this risk in the following ways.
  - We will store all electronic data on a password-protected, encrypted computer.
  - We will keep your identifying information separate from your research data, but we will be able to link it to you. We'll destroy this link after we finish collecting the data.

#### Will there be any cost to me?

There will be no costs to you for participation in this research study.

## Will I be compensated for participating in the study?

For taking part in this research study, you will be paid for your time and inconvenience. After completing the baseline survey, you will be compensated with \$7.00 delivered through the Prolific website. After completing the follow-up survey, available ten weeks after the start of the intervention, you will be compensated \$10.00 through the Prolific website.

# Will my information be confidential?

You will be identified in the research records by a code name or number.

## Will my data be used for future research?

In accordance with scientific norms, the data from this study may be used or shared with other researchers for future research (after removing all personally identifying information).

#### Do I have to participate?

Taking part in this study is voluntary. You are free to not answer any questions or withdraw at any time. Your decision will not change any present or future relationships with Wayne State University or its affiliates.

## Who do I contact if I have questions?

If you have any questions about this study now or in the future, you may contact Halle Thomas or a member of the research team at the following email address: halle.a.thomas@wayne.edu.

This research has been reviewed and approved by an Institutional Review Board (IRB). If you would like to speak with someone other than a member of the research staff, or wish to share feedback privately with the IRB about your research experience, call the Research Participants' Advocate at (313)577-1628 or email <a href="mailto:irbquestions@wayne.edu">irbquestions@wayne.edu</a>. You are encouraged to contact the IRB if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

## **Participation:**

Submission/Revision Date: 2/12/24 Page 2 of 3

Form Date: 12/2023

By completing the baseline survey, you are agreeing to participate in this study. This includes permission to allow researchers to use your data for future research as described in the "Will my data be used for future research" section of this form.

The data that you provide may be collected and used by Qualtrics per its privacy agreement. Additionally, participation in this research is for residents of the United States over the age of 18; if you are not a resident of the United States <u>and/or</u> under the age of 18, please do not complete this survey.

Please save or print a copy of this Information Sheet for your records.

Submission/Revision Date: 2/12/24 Page 3 of 3